CLINICAL TRIAL: NCT07040423
Title: Evaluation of Local Anesthetic Distribution in the PENG Block Compartment Using Pelvic MRI
Brief Title: MRI-Based Assessment of Local Anesthetic Spread in the PENG Block Compartment
Acronym: MRI-PENG
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Campus Bio-Medico University (Other)
Responsible Party: Principal Investigator, Francesca Gargano, Medical doctor, Anesthesiologist, Campus Bio-Medico University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Policlinico Campus Bio-Medico
Record Dates: First submitted 2025-06-10; First posted 2025-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Total Hip Arthroplasty (THA); Postoperative Pain Management After Total Hip Arthroplasty
Keywords: Anesthetics; Anesthetics, Local; Pain; Acute Pain; PENG block; Pelvic MRI; Regional anesthesia; Fascial plane; Local anesthetic spread
MeSH Terms: conditions — Pain; Acute Pain | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PENG Block with MRI-Based Local Anesthetic Spread Assessment (Experimental): All patients receive standardized multimodal analgesia before surgery. Patients in this arm receive an ultrasound-guided PENG block in the supine position under sterile conditions. A low-frequency (2-5 MHz) curvilinear probe is placed above the AIIS and rotated ~45° to align with the pubic ramus. Using an in-plane lateral-to-medial approach, a 10 cm, 20G needle is advanced to the interfascial plane between the iliopsoas tendon and pubic ramus. After negative aspiration, ropivacaine hydrochloride 0.5% is injected in 5 mL increments up to 20 mL, observing spread via ultrasound. A pelvic MRI is then performed to assess anesthetic diffusion before the patient proceeds to total hip arthroplasty.
  Interventions: Procedure: PENG Block; Procedure: Magnetic resonance imaging

INTERVENTIONS:
Procedure: PENG Block — Preoperative ultrasound giuded PENG block (ropivacaine 0,5% 20mL)
Procedure: Magnetic resonance imaging — The patient will undergo a pelvic MRI to assess anesthetic diffusion after PENG block

SUMMARY:
This study uses MRI imaging to evaluate the spread of local anesthetic following the administration of a pericapsular nerve group (PENG) block. The goal is to determine whether a distinct fascial plane exists between neurovascular structures, potentially explaining the block's observed clinical effectiveness.

DETAILED DESCRIPTION:
The pericapsular nerve group (PENG) block has demonstrated promising clinical results in providing analgesia for hip-related pain, particularly in patients with femoral neck fractures or undergoing hip surgery. However, the exact mechanism of action and spread of local anesthetic remain poorly understood. This pilot study aims to use magnetic resonance imaging (MRI) to visualize the distribution pattern of the injectate after PENG block administration.

High-resolution MRI scans will be obtained shortly after the procedure to assess the spatial relationship between the spread of local anesthetic, relevant anatomical structures (including the iliopsoas muscle, femoral artery, and femoral nerve), and potential fascial compartments. The findings will help to clarify the anatomic basis of the PENG block and may guide optimization of technique for enhanced clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for total hip replacement surgery
* Age ≥ 18 years
* ASA physical status classification I-III
* Signed informed consent obtained
* Orthopedic indication for preoperative MRI study

Exclusion Criteria:

* Allergy to local anesthetics
* Infection at the planned puncture site
* Refusal or inability to provide informed consent
* Age < 18 years
* Claustrophobia
* Altered consciousness or severe dementia
* Presence of MRI-incompatible implanted devices (e.g., pacemakers implanted before 2000)
* Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Extent of local anesthetic spread as visualized on MRI after PENG block administration | 10 minutes after injection
  MRI images will be used to assess the diffusion pattern of local anesthetic following PENG (Pericapsular Nerve Group) block. The assessment will focus on whether the anesthetic reaches a specific fascial plane between the femoral vessels and nerves. A radiologist will evaluate the extent and location of the anesthetic spread in relation to key anatomical landmarks (according to centimeter-based measurements as per MRI protocols).

CONTACTS AND LOCATIONS:
Overall Officials: Francesca Gargano, Medical Doctor, Principal Investigator — Policlinico Universitario Campus Bio-Medico
Locations (1):
- Policlinico Universitario Campus Bio-Medico, Roma, Italy, Italy

REFERENCES:
- [Background] Gargano F, Migliorelli S, Pascarella G, Costa F, Strumia A, Bellezze A, Ruggiero A, Carassiti M. A randomized clinical trial comparing different combination of peripheral nerve blocks for intraoperative analgesia in patients on antithrombotic drugs undergoing hip fracture surgery: pericapsular nerve group (PENG) block versus femoral and obturator nerve block. Minerva Anestesiol. 2025 Jun;91(6):524-532. doi: 10.23736/S0375-9393.24.18534-3. Epub 2024 Dec 10. PMID 39656148
- [Background] Nielsen ND, Greher M, Moriggl B, Hoermann R, Nielsen TD, Borglum J, Bendtsen TF. Spread of injectate around hip articular sensory branches of the femoral nerve in cadavers. Acta Anaesthesiol Scand. 2018 Aug;62(7):1001-1006. doi: 10.1111/aas.13122. Epub 2018 Apr 17. PMID 29664158
- [Background] Pascarella G, Costa F, Del Buono R, Pulitano R, Strumia A, Piliego C, De Quattro E, Cataldo R, Agro FE, Carassiti M; collaborators. Impact of the pericapsular nerve group (PENG) block on postoperative analgesia and functional recovery following total hip arthroplasty: a randomised, observer-masked, controlled trial. Anaesthesia. 2021 Nov;76(11):1492-1498. doi: 10.1111/anae.15536. Epub 2021 Jul 1. PMID 34196965
- [Background] Sakamoto J, Manabe Y, Oyamada J, Kataoka H, Nakano J, Saiki K, Okamoto K, Tsurumoto T, Okita M. Anatomical study of the articular branches innervated the hip and knee joint with reference to mechanism of referral pain in hip joint disease patients. Clin Anat. 2018 Jul;31(5):705-709. doi: 10.1002/ca.23077. Epub 2018 Apr 16. PMID 29577432
- [Background] Lee DJ, Elfar JC. Timing of hip fracture surgery in the elderly. Geriatr Orthop Surg Rehabil. 2014 Sep;5(3):138-40. doi: 10.1177/2151458514537273. PMID 25360345